CLINICAL TRIAL: NCT01312454
Title: A Proof of Concept Study to Assess the Safety and IOP-Lowering Effect of AL-59412C Injected Intravitreally
Brief Title: Safety and Intraocular Pressure (IOP) Lowering Effect of AL-59412C
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-10-038
Record Dates: First submitted 2011-03-04; First posted 2011-03-10 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-09

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: intravitreal injection; intraocular pressure; open-angle glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AL-59412C Concentration 1 (Experimental): AL-59412C injectable solution, single intravitreal injection
  Interventions: Drug: AL-59412C injectable solution
- AL-59412C Concentration 2 (Experimental): AL-59412C injectable solution, single intravitreal injection
  Interventions: Drug: AL-59412C injectable solution
- Travoprost (Active Comparator): Travoprost injectable solution, single intravitreal injection
  Interventions: Drug: Travoprost injectable solution
- Vehicle (Placebo Comparator): AL-59412C Vehicle, single intravitreal injection
  Interventions: Drug: AL-59412C Vehicle

INTERVENTIONS:
Drug: AL-59412C injectable solution — Concentration 1 and Concentration 2
  Arms: AL-59412C Concentration 1; AL-59412C Concentration 2
Drug: Travoprost injectable solution
  Arms: Travoprost
Drug: AL-59412C Vehicle — Inactive ingredients used as placebo
  Arms: Vehicle

SUMMARY:
The purpose of this study was to assess the safety and efficacy of AL-59412C injected intravitreally relative to Vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma or ocular hypertension.
* Retinal pathology (eg, retinal degeneration), anterior ischemic optic neuropathy, or vascular occlusion resulting in poor vision in the study eye.
* Able to discontinue all intraocular-lowering (IOP) medications according to the minimum washout period, based upon the class of medication.
* Mean washed out IOP ≥ 24 millimeters mercury (mmHg) to ≤ 36 mmHg at 8 AM in the study eye on two separate Eligibility Visits.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Lens/corneal/vitreal opacity preventing adequate posterior segment visualization of the study eye.
* Current or recent (within 30 days) use of any drug that may prolong the QT interval.
* Poor vision resulting from advanced glaucoma in the study eye.
* Intraocular surgery within the past 6 months in the study eye.
* Ocular laser surgery within the past 3 months in the study eye.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Maximum intraocular (IOP) reduction from baseline up to 24 hours post-injection | Time to event, up to 24 hours post-injection
  IOP was measured by Goldman applanation tonometry at protocol-specified timepoints, up to 24 hours post-injection.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, PhD, Study Director — Alcon Research